CLINICAL TRIAL: NCT02803814
Title: Pancreatoduodenectomy in Pancreatic and Periampullary Tumors: Initial Approach of the Superior Mesenteric Artery Versus Classical Approach: A Prospective, Randomized, Multicenter Study
Brief Title: Pancreatoduodenectomy in Pancreatic and Periampullary Tumors
Acronym: DUOPAN-EPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUOPAN-EPAM
Record Dates: First submitted 2016-05-23; First posted 2016-06-17 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic and Periampullary Tumors
Keywords: Pancreatoduodenectomy; Pancreatic tumors; Periampullary tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superior mesenteric artery approach (Experimental): Initial approach of the superior mesenteric artery to perform a pancreaticoduodenectomy in tumors of the head of the pancreas and peripancreatic area
  Interventions: Procedure: Superior mesenteric artery approach for pancreatoduodenectomy
- Classic approach (Active Comparator): Classic approach to perform a pancreaticoduodenectomy in tumors of the head of the pancreas and peripancreatic area
  Interventions: Procedure: Classic approach for pancreatoduodenectomy

INTERVENTIONS:
Procedure: Superior mesenteric artery approach for pancreatoduodenectomy — Pancreaticoduodenectomy in tumors of the head of the pancreas and peripancreatic area using the superior mesenteric artery approach
  Arms: Superior mesenteric artery approach
Procedure: Classic approach for pancreatoduodenectomy — Pancreaticoduodenectomy in tumors of the head of the pancreas and peripancreatic area using the classical approach
  Arms: Classic approach

SUMMARY:
Background: Recently it has been observed in pancreatic cancer that after apparently complete surgical resection, histological examination of the surgical specimen according to a standard protocol reveals tumor infiltration of the surgical margin in more than 50% of patients. To increase the resection margin and reduce such high infiltration rate, a new surgical approach based on the initial dissection of the superior mesenteric artery has been advocated.

Aims: To compare the rate of free resection margin (R0) and oncological results of two possible approaches to perform a pancreaticoduodenectomy in tumors of the head of the pancreas and peripancreatic area: the classic approach versus the initial approach of the superior mesenteric artery.

Methodology: Prospective, randomized, multicenter study in which patients with pancreatic and periampullary tumors undergo a pancreaticoduodenectomy. In a group the classical approach from the superior mesenteric vein will be performed and in the other group an initially dissecting the superior mesenteric artery approach will be carried out. 116 patients are required and the main variables considered are: free margin rates (R0) or infiltrated by tumor (R1), postoperative morbidity, mortality, local and systemic recurrence, disease-free interval and survival at 1, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic and periampullary tumors undergo a pancreaticoduodenectomy

Exclusion Criteria:

* Patients with hepatic or peritoneal metastasis
* Patients with irresectable tumor
* Patients with R2 resection
* Patients Grade IV of the American Society of Anesthesiology Score
* Patients with neoadjuvant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Rate of free resection margin (R0) | 1 month
  Histological examination of the surgical specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabater L, Cugat E, Serrablo A, Suarez-Artacho G, Diez-Valladares L, Santoyo-Santoyo J, Martin-Perez E, Ausania F, Lopez-Ben S, Jover-Navalon JM, Garces-Albir M, Garcia-Domingo MI, Serradilla M, Perez-Aguirre E, Sanchez-Perez B, Di Martino M, Senra-Del-Rio P, Falgueras-Verdaguer L, Carabias A, Gomez-Mateo MC, Ferrandez A, Dorcaratto D, Munoz-Forner E, Fondevila C, Padillo J. Does the Artery-first Approach Improve the Rate of R0 Resection in Pancreatoduodenectomy?: A Multicenter, Randomized, Controlled Trial. Ann Surg. 2019 Nov;270(5):738-746. doi: 10.1097/SLA.0000000000003535. PMID 31498183